CLINICAL TRIAL: NCT00267592
Title: A Phase II Trial of Talampanel in Conjunction With Radiation Therapy With Concurrent and Adjuvant Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Safety and Efficacy of Talampanel in Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IXR-207-21-189 / NABTT 0304; NCT00082992 (obsolete NCT alias)
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — talampanel; Radiotherapy

ARMS (1):
- enzyme-inducing antiseizure drug (Experimental): A single-arm study with all subjects assigned to one treatment (radiation + temozolomide + talampanel) but subjects receiving concomitant anti-seizure drugs which could increase study drug elimination had a slightly modified dose/schedule of study drug. The primary endpoint is analyzed as a single group.
  Interventions: Drug: Talampanel; Radiation: Radiation Therapy (RT) 5 days a week +; Drug: temozolomide(TMZ) 75mg; Drug: adjuvant TMZ 200mg

INTERVENTIONS:
Drug: Talampanel — Talampanel administered orally TID beginning the first day and continued until there is talampanel-related toxicity or tumor progression.
Radiation: Radiation Therapy (RT) 5 days a week +
Drug: temozolomide(TMZ) 75mg — temozolomide(TMZ) 75mg 3 times daily (TID) for 6 weeks
Drug: adjuvant TMZ 200mg — adjuvant TMZ 200mg TID for 5 consecutive days each month for a total of 6 months.

SUMMARY:
The purpose of this study is to estimate overall survival for adult patients with newly diagnosed glioblastoma multiforme treated with talampanel during radiation therapy with concurrent and adjuvant temozolomide. This study will also determine the toxicity and toxicity rate of talampanel for this therapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age
* Patients must have histologically confirmed supratentorial Grade IV astrocytoma (glioblastoma multiforme)
* Patients must not have prior radiation therapy, chemotherapy (including Gliadel wafer), immunotherapy or therapy with a biologic agent, or hormonal therapy. Glucocorticoid therapy is allowed.
* Patients must have recovered from the immediate post-operative period and be maintained on a stable corticosteroid regimen (on increase for 5 days) prior to the start of treatment.
* Patients must have a Karnofsky performance of at least 60% or more.

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness.
* Patients receiving concurrent chemotherapeutics or investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 24 months

SECONDARY OUTCOMES:
Talampanel-related toxicity | 29 months